CLINICAL TRIAL: NCT05858151
Title: Evaluation of the Transforming Food Systems to Improve Diet Quality and Resilience for the Most Vulnerable Program in Mozambique
Brief Title: Transforming Food System Evaluation in Mozambique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Numbers Whizzy (Unknown); Universidade de Lúrio (Unknown); ANSA (Unknown)
Responsible Party: Principal Investigator, Valerie Flax, Senior Research Public Health Analyst, RTI International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 424601
Record Dates: First submitted 2023-04-19; First posted 2023-05-15 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-07

CONDITIONS: ASF Consumption
Keywords: diet; animal source foods; market intervention; social and behavior change communication intervention; men; women; Mozambique
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Data will be collected through household surveys, market actor surveys and observations, in-depth interviews (IDIs), and focus group discussions (FGDs). The protocol team has selected a subset of the intervention districts for the evaluation and identify an equal number of districts outside the program coverage area with similar characteristics to serve as the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Food system and demand generation
- Control/No Intervention (No Intervention)

INTERVENTIONS:
Behavioral: Food system and demand generation — The Global Alliance for Improved Nutrition (GAIN) will implement the Transforming Food Systems to Improve Diet Quality and Resilience for the Most Vulnerable program, which will use a market-based approach to improving diets through food systems. The set of interventions proposed is based on characteristics and challenges of the food environments of bottom of pyramid consumers in Mozambique. GAIN will focus on elements of the food environment related to accessibility, affordability, and desirability of animal source foods (ASFs) in Mozambique.
  Arms: Intervention

SUMMARY:
Global Alliance for Improved Nutrition (GAIN)'s "Transforming Food Systems to Improve Diet Quality and Resilience for the Most Vulnerable" program seeks to improve consumption of healthy foods by improving supply, increasing demand, and improving the enabling environment for different targeted foods in 4 countries by operating at multiple levels - individuals, households, markets, producers, and policies. RTI and local partners propose to conduct impact and process evaluations of GAIN's program tailored to the theory of change and the target foods for Mozambique. The evaluation in Mozambique will include a mix of quantitative and qualitative methods and will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) implementation research framework.

DETAILED DESCRIPTION:
To increase consumption of animal source foods (ASFs) by Bottom of Pyramid (BoP) consumers, the Global Alliance for Improved Nutrition (GAIN) will implement the Transforming Food Systems to Improve Diet Quality and Resilience for the Most Vulnerable program, which will use a market-based approach to improving diets through food systems. The set of interventions proposed is based on characteristics and challenges of the food environments of bottom of BoP consumers in Mozambique. GAIN will focus on elements of the food environment related to accessibility, affordability, and desirability of animal source foods (ASFs) in Mozambique.

GAIN's program will improve accessibility (physical distance that consumers travel to procure food) by developing sustainable last mile ASF delivery systems. This will involve developing an efficient and integrated private sector-led delivery system of fish (fresh and dry), chicken cuts (tails, heads, feet, necks, guts), and eggs from consolidation points/aggregators to last-mile retailers by facilitating logistics services (including on-demand backhaul trucks) and strengthening the linkages along the ASF supply chain. Accessibility will also be increased through improvement of fish drying technology and practices using solar tent dryers to enhance the quality and shelf life of dried fish, improve food safety, and decrease salt content.

GAIN intends to improve affordability of ASF by focusing on improving the value chains of the most affordable ASF options (fish, chicken cuts, and eggs) and will support accessibility by investing in enhanced cold chain systems and stronger distribution channels to underserved areas.

GAIN's program will improve desirability through a demand generation campaign to increase the frequency of ASF consumption among BoP consumers by focusing on key messages that are expected to drive behavior change. The campaign will focus on promoting ASFs as a food group for the whole family, using a short and catchy slogan. Messages will be disseminated through provincial and community radio via drama-based radio messages with new spots every 2 weeks, a musical jingle, and interactive call-in shows. Complementary channels will include television (cooking shows showing preparation of promoted foods), radio messages, social media campaigns, and illustrative point of sale materials (e.g., posters, danglers).

This evaluation of GAIN's Transforming Food Systems to Improve Diet Quality and Resilience for the Most Vulnerable program in Mozambique will use a mixed-methods quasi-experimental parallel group before-after cross-sectional design to assess effectiveness on increasing frequency of animal source food (ASF) consumption by bottom of the pyramid (BoP) consumers. The evaluation will be carried out in 4 intervention and 4 comparison districts, purposefully selected. It will include both impact and process evaluation components. Data will be collected through household surveys, market actor surveys and observations, in-depth interviews (IDIs), and focus group discussions (FGDs). Cross-sectional population-based household surveys with men and women in BoP households will be conducted at baseline (N=1,472) and endline (N=1,472) to assess the impact of the intervention on their ASF consumption frequency and dietary diversity using difference-in-differences analysis. Market actor surveys and observations will be conducted with retailers of fish, chicken, and eggs in both study arms at baseline and endline (N=800 at each time point). The baseline-endline market actor data will be analyzed using difference-in-difference analysis to assess improvements in availability, food safety, and prices of fish, chicken, and eggs. Process evaluation data will include IDIs with food transporters, traders, large-scale retailers, and other stakeholders (N=16 at each timepoint); FGDs with retailers of the target foods (N=16 FGDs at each time point); and FGDs with BoP households (N=16 FGDs at each time point). These will be conducted at midline and endline in the intervention districts only. Qualitative data will be analyzed using thematic content analysis methods. We will link the process and impact data through a program impact pathway analysis to document the pathways through which the program achieved its effects.

ELIGIBILITY:
Household Surveys

Inclusion Criteria:

* Reside in the enumeration areas;
* Be a man ≥ 18 years or a woman 18-49 years;
* The household earns <$3.20 per person per day;
* Be able to speak one of the main local languages and/or Portuguese;
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Have a mental or psychological illness that prevents them from understanding the study;
* Have any physical illness that prevents them from being safely and constructively involved in the investigation;
* Be under the age of 18 years at the time of the study.

Market Actor Surveys

Inclusion Criteria:

* Be a retailer of fish, chicken or eggs in one of the markets in the districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Portuguese;
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Have a mental or psychological illness that prevents them from understanding the study;
* Have any physical illness that prevents them from being safely and constructively involved in the investigation;
* Be under the age of 18 years at the time of the study.

In-depth interviews with market actors:

Inclusion criteria:

* Be a food transporter, trader, large-scale retailer, government official or other stakeholder involved in market-related activities in the fish, chicken or egg value chains in the intervention districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Portuguese;
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Have any mental or psychological illness that prevents them from understanding the study
* Have any physical illness that prevents them from being safely and constructively involved in an investigation;
* Be under the age of 18 at the time of the study.

Focus group discussion (FGD) participants will be selected from lists of participants in the market actor and household surveys and will be consented again for the FGDs if they meet the following criteria:

FGDs) with market actors:

Inclusion criteria:

* Be a small-scale retailer of fish, chicken, or eggs in intervention districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Portuguese;
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Have any mental or psychological illness that prevents them from understanding the study;
* Have any physical illness that prevents them from being safely and constructively involved in an investigation;
* Be under the age of 18 at the time of the study.

FGDsocus group discussions with households:

Inclusion criteria:

* Belong to a BoP household living in a community in the intervention districts selected for the evaluation;
* Be over 18 years old;
* Be able to speak one of the main local languages and/or Portuguese;
* Provide informed consent to participate in the study.

Exclusion Criteria:

* Have any mental or psychological illness that prevents them from understanding the study
* Have any physical illness that prevents them from being safely and constructively involved in an investigation;
* Be under the age of 18 at the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5216 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
ASF frequency of consumption | Baseline (May 2023), endline (May 2026 (3 years))
  Change in the mean frequency of fish, chicken, and egg consumption during the last 7 days by men and women in BoP households

SECONDARY OUTCOMES:
Percent of household members with increased knowledge of target ASFs | Baseline (May 2023), endline (May 2026 (3 years))
  Percent of household members

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Costa, Principal Investigator — Universidade Lúrio
Locations (1):
- Numbers Whizzy, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be shared through Nesstar